CLINICAL TRIAL: NCT06142877
Title: Identifying and Addressing the Effects of Social Media Use on Young Adults' E-Cigarette Use: A Solutions-Oriented Approach
Brief Title: Effects of Social Media Use on Young Adults' E-Cigarette Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Stanford University (Other); University of Southern California (Other); University of Wisconsin, Madison (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15427; K01DA055073 (NIH)
Record Dates: First submitted 2023-11-15; First posted 2023-11-22 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Electronic Cigarette Use
Keywords: social media; young adult; e-cigarette; nicotine vaping
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two groups: 1) social media use reduction (intervention), or 2) social media use as usual (control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Media Use Reduction (Experimental)
  Interventions: Behavioral: Social Media Use Reduction
- Social Media Use as Usual (No Intervention)

INTERVENTIONS:
Behavioral: Social Media Use Reduction — Participants will be incentivized to reduce their social media use by a pre-specified percentage from baseline.
  Arms: Social Media Use Reduction

SUMMARY:
The goal of this clinical trial is to test the effects of social media use on e-cigarette use in young adults who use e-cigarettes. The main questions it aims to answer are:

* Does reducing social media use change young adults' e-cigarette use?
* Does reducing social media use change things such as young adults' mental health and what they see on social media?

Participants will complete surveys and submit screenshots showing how much time they spend on social media.

Researchers will compare young adults who reduce their social media use to young adults who use social media as usual, to see if their e-cigarette use differs.

DETAILED DESCRIPTION:
The overall goals of this project are to understand how young adults' social media use affects their nicotine vaping and to identify intervention targets that mitigate social media's impact on vaping. Prevalence of vaping and social media use among young adults have increased in tandem. Exposure to vaping-related social media content is common and is associated with vaping. Intense social media use appears to contribute to young adults' increased mental health symptoms, which are linked to tobacco product use. This project aims to contribute to scientific understanding of the causal links between social media use and vaping in young adulthood. Young adults with past-month vaping will report time spent on social media, vaping-related social media content exposure, social comparison on social media, mental health, and vaping behavior. After a 1-month baseline measurement period, they will be randomized to reduce their social media use (incentivized) or use social media as usual for a 3-month experimental period. Longitudinal within- and between-subjects analyses will test relationships between time spent on social media, risk factors for vaping, and vaping behavior. Specific research aims are to: (1) investigate the relationships between a reduction in social media use and: a) vaping content exposure, b) social comparison, and c) mental health, and (2) examine whether reducing social media use reduces past-month vaping days, vaping episodes per vaping day, and puffs per vaping episode.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-25
* Daily social media use
* Ownership of a smartphone
* Vaping (i.e., use of a nicotine e-cigarette) on 1-19 days of the past 30 days
* Residing in the United States

Exclusion Criteria:

-Lack of capacity to provide informed consent

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Past-month vaping days | Collected at baseline, 1mo, 3mo, 6mo
  Number of days the participant vaped nicotine in the past 30 days

SECONDARY OUTCOMES:
Episodes per vaping day | Collected at baseline, 1mo, 3mo, 6mo
  Average number of times the participant used a nicotine vaping device on each day (of the past 30) they vaped nicotine
Puffs per vaping episode | Collected at baseline, 1mo, 3mo, 6mo
  Past-month number of puffs per nicotine vaping episode (1-20)

CONTACTS AND LOCATIONS:
Overall Officials: Erin A Vogel, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data will be available from the Principal Investigator upon reasonable request.